CLINICAL TRIAL: NCT00608374
Title: A Randomised Trial of Chlorambucil Versus Fludarabine as Initial Therapy of Waldenström's Macroglobulinaemia and Splenic Lymphoma With Villous Lymphocytes
Brief Title: Chlorambucil or Fludarabine as First-Line Therapy in Treating Patients With Previously Untreated Waldenström Macroglobulinemia, Splenic Lymphoma, or Lymphoplasmacytic Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taunton and Somerset Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000581143; TSH-WM1; ISRCTN56052618
Record Dates: First submitted 2007-12-21; First posted 2008-02-06 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia; splenic marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — Chlorambucil; fludarabine phosphate

INTERVENTIONS:
Drug: chlorambucil
Drug: fludarabine phosphate
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as chlorambucil and fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known whether chlorambucil is more effective than fludarabine in treating Waldenström macroglobulinemia, splenic lymphoma, or lymphoplasmacytic lymphoma.

PURPOSE: This randomized phase III trial is studying chlorambucil to see how well it works compared with fludarabine as first-line therapy in treating patients with previously untreated Waldenström macroglobulinemia, splenic lymphoma, or lymphoplasmacytic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of first-line therapy comprising chlorambucil vs fludarabine phosphate in patients with previously untreated Waldenström macroglobulinemia, splenic lymphoma with villous lymphocytes, or non-IgM lymphoplasmacytic lymphoma.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (Waldenström macroglobulinemia vs splenic lymphoma with villous lymphocytes vs non-IgM lymphoplasmacytic lymphoma). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral chlorambucil on days 1-10. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive fludarabine phosphate orally or IV on days 1-5. Treatment repeats every 28 days for 3-6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo quality of life assessment at baseline.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Waldenström macroglobulinemia, splenic lymphoma with villous lymphocytes (SLVL), or non-IgM lymphoplasmacytic lymphoma based on morphological and immunophenotypic criteria

  * Bone marrow should be assessed by two-color flow cytometry for the expression of the following antigens:

    * Surface Ig
    * CD19
    * CD20
    * CD5
    * CD10
    * CD23
* Previously untreated disease requiring therapeutic intervention (as judged by the primary physician), as indicated by ≥ 1 of the following:

  * Hemoglobin < 10 g/dL
  * ANC < 1.5 x 10^9/L
  * Platelet count < 150 x 10^9/L
  * Clinical evidence of hyperviscosity in terms of neurological or ocular disturbance
* Patients with disease detected by clonal cells alone are not eligible

PATIENT CHARACTERISTICS:

* Performance status 0-2
* Life expectancy > 6 months
* Serum creatinine < 200 mmol/L
* AST and ALT < 2 times upper limit of normal
* Negative direct Coomb's test
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* No severe or life-threatening cardiac, pulmonary, neurological, psychiatric, or metabolic disease
* No other concurrent malignancy
* No AIDS or AIDS-related complex
* No evidence of active hepatitis C infection

PRIOR CONCURRENT THERAPY:

* Prior plasmapheresis for control of clinically significant hyperviscosity allowed
* Prior splenectomy for SLVL allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Response to therapy (complete and partial response rates)
Duration of response

SECONDARY OUTCOMES:
Improvement in hematological parameters
Toxicity
Quality of life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life-30 questionnaire
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Roger G. Owen, MD, MRCP, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (49):
- Australia (5):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
- United Kingdom (44):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - North Devon District Hospital, Barnstaple, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Royal United Hospital, Bath, England
  - City Hospital - Birmingham, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bradford Royal Infirmary, Bradford, England
  - Queen's Hospital, Burton-on-Trent, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Saint Richards Hospital, Chichester, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Russells Hall Hospital, Dudley, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Harrogate District Hospital, Harrogate, England
  - Hereford Hospitals, Hereford, England
  - Watford General Hospital, Herts, England
  - Wycombe General Hospital, High Wycombe, England
  - Hull Royal Infirmary, Hull, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Leeds General Infirmary, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - University College Hospital - London, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Trafford General Hospital, Manchester, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Derriford Hospital, Plymouth, England
  - Pontefract General Infirmary, Pontefract West Yorkshire, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Rotherham General Hospital, Rotherham, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Staffordshire General Hospital, Stafford, England
  - Taunton and Somerset Hospital, Taunton Somerset, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Kent and Sussex Hospital, Tunbridge Wells, Kent, England
  - Sandwell General Hospital, West Bromwich, England
  - New Cross Hospital, Wolverhampton, England
  - Monklands General Hospital, Airdrie, Scotland
  - Southern General Hospital, Glasgow, Scotland
  - Pinderfields General Hospital, Wakefield, Scotland
  - Ysbyty Gwynedd, Bangor, Wales

REFERENCES:
- [Derived] Leblond V, Johnson S, Chevret S, Copplestone A, Rule S, Tournilhac O, Seymour JF, Patmore RD, Wright D, Morel P, Dilhuydy MS, Willoughby S, Dartigeas C, Malphettes M, Royer B, Ewings M, Pratt G, Lejeune J, Nguyen-Khac F, Choquet S, Owen RG. Results of a randomized trial of chlorambucil versus fludarabine for patients with untreated Waldenstrom macroglobulinemia, marginal zone lymphoma, or lymphoplasmacytic lymphoma. J Clin Oncol. 2013 Jan 20;31(3):301-7. doi: 10.1200/JCO.2012.44.7920. Epub 2012 Dec 10. PMID 23233721
- [Derived] Nguyen-Khac F, Lambert J, Chapiro E, Grelier A, Mould S, Barin C, Daudignon A, Gachard N, Struski S, Henry C, Penther D, Mossafa H, Andrieux J, Eclache V, Bilhou-Nabera C, Luquet I, Terre C, Baranger L, Mugneret F, Chiesa J, Mozziconacci MJ, Callet-Bauchu E, Veronese L, Blons H, Owen R, Lejeune J, Chevret S, Merle-Beral H, Leblondon V; Groupe Francais d'Etude de la Leucemie Lymphoide Chronique et Maladie de Waldenstrom (GFCLL/MW); Groupe Ouest-Est d'etude des Leucemie Aigues et Autres Maladies du Sang (GOELAMS); Groupe d'Etude des Lymphomes de l'Adulte (GELA). Chromosomal aberrations and their prognostic value in a series of 174 untreated patients with Waldenstrom's macroglobulinemia. Haematologica. 2013 Apr;98(4):649-54. doi: 10.3324/haematol.2012.070458. Epub 2012 Oct 12. PMID 23065509